CLINICAL TRIAL: NCT03552991
Title: Effects of Dietary Fiber on Glucose Control in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Bukwang Pharmaceutical, Co., Ltd. (Industry); ChunLab, Inc. (Unknown)
Responsible Party: Principal Investigator, MOON-KYU LEE, Professor, Division of Endocrinology and Metabolism, Department of Internal Medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Agio study
Record Dates: First submitted 2018-05-17; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Dietary Fiber; Microbiota; Diabetes Mellitus, Type 2; Metformin; Sulfonylurea Compounds
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Agio arm (Other): It is a pilot study based on the proof-of-concept that dietary fiber helps glucose control in patients with type 2 diabetes. As a single-arm study, 'Agiocur Pregranules' (dietary fiber) is administered for 28 days and stopped for next 28 days, in patients with type 2 diabetes.
  Interventions: Drug: Agiocur Pregranules

INTERVENTIONS:
Drug: Agiocur Pregranules — 6g before breakfast and 12g after dinner for first 28 days, and no medication for next 28 days for washout
  Other Names: Agio gran.

SUMMARY:
The purpose of this study is to determine the effect of a commercial dietary fiber supplement on patients with type 2 diabetes mellitus, in the way of glucose control, insulin action in the body, and the gut microbiota (bacteria) abundance.

DETAILED DESCRIPTION:
Fiber supplements such as psyllium are known to be beneficial to glycemic control in patients with type 2 diabetes mellitus (T2DM). Gut microbiota has a role in regulating host energy metabolism and systemic inflammation by several pathways such as short-chain fatty acid production, fasting-induced adipose factor expression, endocannabinoid system, and gut epithelial permeability. As dietary components can influence the composition of the microbiota, we hypothesized that fiber supplements could modify gut microbiota and consequently affect glycemic control and inflammatory condition in patients with T2DM.

The primary outcome was to assess the effect of fiber on glucose control (by comparing fasting glucose and glycoalbumin), insulin secretion and sensitivity. Secondary outcomes were the changes abundance of microbiota, incretins, and lipopolysaccharide (LPS).

ELIGIBILITY:
Inclusion Criteria (all of the followings):

* Among type 2 diabetic patients who visit Diabetes Center at Samsung Medical Center
* 2 or more of following are required:

  1. use of lipid-lowering drugs and / or triglyceride ≥ 150 mg/dL, high-density lipoprotein < 40 mg/dL in men and < 50 mg/dL in women
  2. waist circumference > 90 cm in men and > 80 cm in women
  3. antihypertensive medication and / or blood pressure ≥ 130/85 mmHg
* Hemoglobin A1c level 7.0 - 9.0% (6.5 - 9.0% in age 50-60 years old)
* Patients who are treated with combination therapy of sulfonylurea and metformin at least 6 months and in steady-glucose-controlled state.

Exclusion Criteria (at least one of the followings):

* Patients using insulin, alpha-glucosidase inhibitor, meglitinide, thiazolidinedione, or incretin agent (both oral or injectables)
* Recently diagnosed (within 6 months) acute diabetic complication such as diabetic ketoacidosis and hyperosmolar hyperglycemic state
* Clinically significant cardiovascular disease
* Patients treated with oral or intravenous antibiotics last 12 months
* Patients who took fiber supplements last 6 months
* Fasting serum c-peptide level < 1 ng/mL
* Duration of type 2 diabetes > 10 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Glycoalbumin | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Insulinogenic index | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Quantitative insulin sensitivity check index (QUICKI) | the 4th week of study
  By comparing the level of 4th week, compared to baseline. QUICKI is derived from fasting blood glucose and insulin level, reflecting insulin sensitivity.

SECONDARY OUTCOMES:
Microbiota composition change | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Incretins (GIP) | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Incretins (GLP-1) | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Incretins (GLP-2) | the 4th week of study
  By comparing the level of 4th week, compared to baseline
Lipopolysaccharide (LPS) | the 4th week of study
  By comparing the level of 4th week, compared to baseline

REFERENCES:
- [Result] Kim DJ. The epidemiology of diabetes in Korea. Diabetes Metab J. 2011 Aug;35(4):303-8. doi: 10.4093/dmj.2011.35.4.303. Epub 2011 Aug 31. PMID 21977448
- [Result] Kim JH, Kim DJ, Jang HC, Choi SH. Epidemiology of micro- and macrovascular complications of type 2 diabetes in Korea. Diabetes Metab J. 2011 Dec;35(6):571-7. doi: 10.4093/dmj.2011.35.6.571. Epub 2011 Dec 26. PMID 22247898
- [Result] Slavin JL. Position of the American Dietetic Association: health implications of dietary fiber. J Am Diet Assoc. 2008 Oct;108(10):1716-31. doi: 10.1016/j.jada.2008.08.007. PMID 18953766
- [Result] Bajorek SA, Morello CM. Effects of dietary fiber and low glycemic index diet on glucose control in subjects with type 2 diabetes mellitus. Ann Pharmacother. 2010 Nov;44(11):1786-92. doi: 10.1345/aph.1P347. Epub 2010 Oct 19. PMID 20959501
- [Result] Burcelin R, Serino M, Chabo C, Blasco-Baque V, Amar J. Gut microbiota and diabetes: from pathogenesis to therapeutic perspective. Acta Diabetol. 2011 Dec;48(4):257-273. doi: 10.1007/s00592-011-0333-6. Epub 2011 Oct 2. PMID 21964884
- [Result] Walker AW, Ince J, Duncan SH, Webster LM, Holtrop G, Ze X, Brown D, Stares MD, Scott P, Bergerat A, Louis P, McIntosh F, Johnstone AM, Lobley GE, Parkhill J, Flint HJ. Dominant and diet-responsive groups of bacteria within the human colonic microbiota. ISME J. 2011 Feb;5(2):220-30. doi: 10.1038/ismej.2010.118. Epub 2010 Aug 5. PMID 20686513
- [Result] Maslowski KM, Mackay CR. Diet, gut microbiota and immune responses. Nat Immunol. 2011 Jan;12(1):5-9. doi: 10.1038/ni0111-5. PMID 21169997